CLINICAL TRIAL: NCT06212375
Title: Vegetable Offering in the Home Environment - Impact of Free Accessibility and Choice on Snack Vegetable Intake
Acronym: VOHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Collaborators: OnePlanet Research Center Wageningen (Unknown)
Responsible Party: Principal Investigator, Marlou Lasschuijt, Dr. Marlou Lasscuijt, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: VOHEStudy
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Within subject study design: All children receive the four possible combinations of interventions.
  Interventions: Behavioral: Vegetable variety; Behavioral: Vegetable offering strategy

INTERVENTIONS:
Behavioral: Vegetable variety — Either children are offered a variety of three vegetables or a single vegetable.
Behavioral: Vegetable offering strategy — Either children can decide when to eat their vegetables or parents initiate a moment.

SUMMARY:
This study examines the impact of offering strategies on the fruit and vegetable intake of children aged 4-6. Two key factors being explored are whether caregivers initiate the offering or if it's freely provided and whether children have a choice in selecting fruits and vegetables. The objective is to determine how these strategies affect the children's fruit and vegetable intake.

The research follows a 2x2 factorial cross-over design, with participants exposed to four different conditions. Interventions involve home visits, informed consent, questionnaires, and children tasting vegetables to assess their preferences. A SnackBox is placed in the home, and parents ensure it's filled based on the condition - children either choose a snack vegetable or have it initiated by parents. Daily questionnaires about vegetable consumption are completed, and the study concludes with material collection.

The study includes 44 children aged 4-6 and carries minimal risks with no immediate benefits. Caregivers spend around four hours participating in the study.

DETAILED DESCRIPTION:
Rationale: The dietary habits formed during early childhood play a pivotal role in shaping long-term health outcomes. Adequate consumption of fruits and vegetables during this critical developmental period is associated with reduced risk of chronic diseases and the promotion of overall well-being. However, achieving optimal fruit and vegetable intake in young children can be challenging, and understanding the influence of offering strategies on their dietary choices is of paramount importance. The present study aims to investigate the effect of offering strategy on the fruit and vegetable intake of children aged 4-6 years old. Specifically, we will explore two key dimensions of offering strategy: (1) whether the offering is freely provided or initiated by caregivers and (2) whether children are given a choice or not in their selection of fruits and vegetables. These factors have the potential to significantly impact children's dietary behaviors.

Objective: To determine the effect of offering strategy (freely offered vs initiated and choice vs no-choice) on fruit and vegetable intake (gram) of children aged 4-6 years old.

Study design: The study will follow a 2 ((freely offered vs initiated) x 2 (choice vs no-choice) factorial cross-over design. Participants are exposed, in duplicate, to each of the four condition combinations.

Interventions: The research team visits the participants at home for an intake session, during which parents provide informed consent, complete questionnaires, and children taste the vegetables to assess their liking. During the measurement afternoons, a SnackBox is placed in the home environment, and parents ensure it is filled. Depending on the condition, parents either allow children to freely take a snack vegetable or initiate when they can eat them. Three vegetables (carrots, bell peppers, cucumbers) are offered in the choice condition, while only one vegetable is available in the no-choice condition. Parents are notified to complete a daily questionnaire about vegetable consumption during dinner at the end of each day. The research team returns to collect all study materials, concluding the study.

Study population: 44 children between 4 to 6 years old. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study is non-therapeutic to the subjects. No immediate benefits for the subjects are expected from participation in this study, and the risk associated with participation can be considered negligible. In terms of time, the subject's burden is as follows: 1 hour for the intake session and corresponding questionnaires prior to the intervention sessions for the caregiver and 15 minutes for the child; 8 times 20 minutes for completing the daily questionnaires and serving vegetables and lastly for the parent and child, 20 minutes for the wrap-up session after the intervention period. This results in a total of 4 hours for the caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Children should be between 4-7 years old;
* Children should spend 2 out of 5 afternoons at home on school days, while there is also a caregiver present to offer the vegetables;
* Both caregivers as well as the child are willing to comply to the study procedure;

Exclusion Criteria:

* Children who have any allergies or intolerances to the fruits and vegetables used in the study;
* Not willing to eat the test foods because of eating habits or beliefs as indicated by parent or caregiver;

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
consumption during the measurement afternoons | 8 afternoons as chosen by the participant
  Consumption during each of the measurement afternoons is measured using the SnackBox. The SnackBox assumes consumption when decreases in weight are detected. To assess the effect of both offering strategies and there interaction, a two-way ANOVA is conducted.

SECONDARY OUTCOMES:
true consumption | 8 afternoons as chosen by the participant
  the weight of the three study-foods is measured before and after the study period is measured and additionally bought foods are registered. Pre-study weight + additionally bought foods - Post-study weight = total true consumption. The SnackBox uses an algorithm to detect decreases in weight and assumes these are due to consumption of snack vegetables. Summation of these decreases in weight results in total consumption measured by the SnackBox. Total true consumption is compared to the SnackBox measured consumption using a Bland-Altman plot and by calculating the Intra Class Correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No